CLINICAL TRIAL: NCT03952065
Title: A Phase II/III Randomized Trial of Comparison of Survival Benefit of Administration of PD1/PDL1/CTLA4 Inhibitors or Their Combinations Via Neck Artery or Intratumor Versus Vein Infusion for Immunotherapy of HNC
Brief Title: IT or IA Infusion of PD1/PDL1/CTLA4 Inhibitors Versus IV for Immunotherapy of Head/Neck Cancers (HNC)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZZITICI-009
Record Dates: First submitted 2019-05-13; First posted 2019-05-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Head/Neck Neoplasm
Keywords: Head/Neck tumor; PD1 antibody; Artery infusion; PDL1 antibody; CTLA4 antibody; Intra-tumor; Interventional therapy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD1/PDL1/CTLA4 inhibitor or their combinations infusion via neck artery (Experimental): Interventional technique is used to localize neck artery to infuse the inhibitor or their combinations directly into tumor.
  Interventions: Drug: PD1/PDL1/CTLA4 inhibitors
- PD1/PDL1/CTLA4 inhibitor or their combinations infusion via peripheral vein (Experimental): Routine peripheral vein infusion of PD1/PDL1/CTLA4 inhibitor or their combinations is performed.
  Interventions: Drug: PD1/PDL1/CTLA4 inhibitors
- PD1/PDL1/CTLA4 inhibitor or their combinations infusion via intra-tumor penetration (Experimental): Interventional technique is used to intra-tumor injection of the inhibitor or their combinations directly into tumor.
  Interventions: Drug: PD1/PDL1/CTLA4 inhibitors

INTERVENTIONS:
Drug: PD1/PDL1/CTLA4 inhibitors — Infusion of PD1/PDL1/CTLA4 inhibitors through peripheral vein or neck artery/intra-tumor.

SUMMARY:
This trial was designed to investigate the survival outcomes, response rates, and safety of patients with advanced Head/Neck Squamous cancer via intra-tumor or intra-artery versus vein infusion of PD1/PDL1/CTLA4 inhibitor or their combinations.

DETAILED DESCRIPTION:
Head/Neck cancer is a kind of hard-to-treat malignancy worldwide and its overall survival rate is still low. PD1/PDL1/CTLA4 inhibitors are widely used to treat various of cancers now. Delivery of antibody drugs through interventional approaches including intra-tumor or intra-artery, based on the theory of "first pass effect" of drug, can significantly increase the local drug concentration of the tumor, improve the efficacy, and reduce systemic adverse reactions.

To the investigator's knowledge, no studies have been developed on the survival benefit of neck artery infusion or intra-tumor injection of immunotherapeutic agents in patients with advanced HNC. This phase II-III clinical trial was designed to compare the effects of PD1/PDL1/CTLA4 inhibitor or their combinations via IA/IT and IV on the survival benefit of patients with advanced HNC, including ORR, DCR, median survival time, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Cytohistological confirmation is required for diagnosis of HNC.
2. Signed informed consent before recruiting.
3. Age between 18 to 80 years with estimated survival over 3 months.
4. ECOG score < 2
5. Tolerable coagulation function or reversible coagulation disorders
6. Laboratory examination test within 7 days prior to procedure: WBC≥3.0×10E9/L; Hb≥90g/L； PLT ≥50×10E9/L；INR < 2.3 or PT < 6 seconds above control；Cr ≤ 145.5 umul/L；Albumin > 28 g/L；Total bilirubin < 51 μmol/L
7. At least one tumor lesion meeting measurable disease criteria as determined by RECIST v1.1.
8. Patients with advanced HNC which would not be suitable for treatment with loco-regional therapies or have progressed following locoregional therapy such as surgical resection and other treatment.
9. Birth control.
10. Willing and able to comply with scheduled visits, treatment plan and laboratory tests.

Exclusion Criteria:

1. Patients participated in other clinical trials of equipment or drugs (signed informed consent) within 4 weeks;
2. Any serious accompanying disease, which is expected to have an unknown, impact on the prognosis, include heart disease, inadequately controlled diabetes and psychiatric disorders;
3. Patients accompanied with other tumors or past medical history of malignancy;
4. Pregnant or lactating patients, all patients participating in this trial must adopt appropriate birth control measures during treatment;
5. Patients have poor compliance.

   Any contraindications for neck artery infusion procedure:

   A. Impaired clotting test (platelet count < 60000/mm3, prothrombin activity < 50%).

   B. Renal failure / insufficiency requiring hemo-or peritoneal dialysis. C. Known severe atheromatosis. D. Known uncontrolled blood hypertension (> 160/100 mm/Hg).
6. Allergic to adriamycin chemotherapy drugs，contrast agent or lipiodol;
7. Any agents which could affect the absorption or pharmacokinetics of the study drugs
8. Subjects unable to suffer the discomfort of the artery infusion procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Overall survival (OS) will be defined as the elapsed time from the enrollment to death from any cause. For surviving patients, follow-up will be censored at the date of last contact (or last date known to be alive). Follow-up for OS will occur every 12 weeks (±1 month) until death or withdrawal of consent from the study.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  Progression-free survival (PFS) will be defined as the elapsed time from the first date of study treatment until documented disease progression (as per mRECIST) or death from any cause, whichever is earlier. For patients who remain alive without progression, follow-up time will be censored at the date of last disease assessment.
Adverse event rate | 2 years
  Adverse event rate will be defined as the rate of patients who developed adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Lian, MD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University; Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guanzhou, Guangdong, China